CLINICAL TRIAL: NCT00388336
Title: A Pilot Study to Evaluate the Response Rate of PROCRIT� (Epoetin Alfa) at 60,000 Units Every Two Weeks in Anemic Cancer Patients Not Receiving Chemotherapy Or Radiation Therapy
Brief Title: PROCRIT (Epoetin Alfa) 60,000 Units Administered Once Every Two Weeks in Anemic Cancer Patients Who Are Not Receiving Chemotherapy or Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004594; NCT00090935 (obsolete NCT alias)
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Neoplasms
Keywords: Anemia; Neoplasms, Hemoglobin values; PROCRIT; Epoetin alfa
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin Alfa

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of Epoetin alfa administered at 60,000 Units every two weeks in cancer patients who are not receiving chemotherapy or radiation therapy.

DETAILED DESCRIPTION:
This was an open-label (doctors and patients knew which drug was being administered), non-randomized (patients were assigned to treatment), multi-center pilot study with the objective to investigate the effectiveness of PROCRIT (Epoetin alfa) on hematopoietic response (effect on red blood cells) when administered at 60,000 Units subcutaneously (under the skin) every two weeks in anemic patients with cancer who were not receiving chemotherapy or radiation therapy.

Treatment with study drug was for a maximum of 12 weeks followed by a 4-week observation period after the last dose of the study drug had been administered.

Safety and efficacy evaluations were performed at specified intervals throughout the study and included assessment of laboratory tests (Complete Blood Count [CBC], Serum Chemistry [including hemoglobin level]), vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events. All patients enrolled in this study received pharmacologic ferrous sulfate 325 mg by mouth once a day or an equivalent formulation, as tolerated, unless it was determined by the physician that the patient should not receive it. All patient's received injections of PROCRIT (Epoetin alfa) 60,000 Units under the skin once every two weeks. If after 4 weeks of treatment, the patient's hemoglobin level did not increase by >= 1 g/dL, the Epoetin alfa dose was increased to 80,000 Units every 2 weeks. Study drug was administered for a maximum of 12 weeks followed by a 4-week observation period after the last dose of study drug. Epoetin alfa doses were reduced or held as needed depending on the patients' hemoglobin level.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of non-myeloid malignancy
* Baseline hemoglobin value of <= 11 g/dL unrelated to transfusion
* Patients must not be receiving or planning to receive chemotherapy or radiotherapy within the 16-week study period. However, patients receiving hormonal therapy or non-myelosuppressive therapies are allowable
* Female patients with reproductive potential must have a negative serum pregnancy test at screening.

Exclusion Criteria:

* Patients must not have uncontrolled hypertension or a history (within 6 months) of uncontrolled cardiac arrhythmias, pulmonary emboli, deep vein thrombosis, ischemic stroke, other arterial or venous thrombotic events (excluding superficial thromboses), or known history of chronic coagulation disorder
* No transfusion within 28 days prior to first dose
* No planned chemotherapy or radiation during study and no prior chemotherapy within 8 weeks or radiation within 4 weeks of study entry
* No prior treatment with Epoetin alfa or any other erythropoietic agent within the previous two months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-02; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was to evaluate hematopoietic response, defined as >= 2 g/dL Hb increase from baseline and/or Hb >= 12 g/dL over the course of the study and independent of transfusion within 28 days.

SECONDARY OUTCOMES:
Secondary endpoints included the effects of PROCRIT (Epoetin alfa) on transfusion requirements, on Quality of Life as measured by the Linear Analog Scale Assessment (LASA) and FACT-An tools as well as time to hemoglobin response.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Pilot Study to Evaluate the Response Rate of PROCRIT (Epoetin Alfa) at 60,000 Units Every Two Weeks in Anemic Patients with Cancer Not Receiving Chemotherapy or Radiation Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=602&filename=CR004594_CSR.pdf